CLINICAL TRIAL: NCT07002125
Title: The Effect of Whole Body Vibration Therapy on Muscle Oxygenation in Individuals With Type 2 Diabetes: A Randomized Controlled Trial
Brief Title: Whole Body Vibration Therapy in Individuals With Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Medipol University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Selcan Suicmez, Principal Investigator, Ankara Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GaziU-FTR-SS-02
Record Dates: First submitted 2025-05-17; First posted 2025-06-03 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes; Whole Body Vibration; Muscle Oxygenation; Aerobic Exercise
Keywords: Aerobic exercise; diapason; balance; HbA1c; type 2 diabetes; whole body vibration; muscle oxygenation
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Individuals with Type 2 diabetes who agreed to participate in the study will be divided into two groups as aerobic exercise group (AE) and whole body vibration group (AE+WBV).
Who Masked: Participant, Outcomes Assessor
Masking Description: The study is planned as a triple-blind, randomized controlled trial. Patients will not be informed about their group. The assessment will be followed by 1 physiotherapist, and the exercise program will be followed by 2 physiotherapists (the physiotherapist performing the assessment is not included). Study groups will be coded before statistical analysis, and the meaning of the codes will not be told to the statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise (Experimental): The aerobic exercise group (AE) will participate in an ascending aerobic exercise program for 8 weeks, 3 sessions per week.
  Interventions: Other: Aerobic Exercise
- Whole Body Vibration (Experimental): The whole body vibration group (AE+TVV) will additionally participate in an 8-week incremental aerobic exercise program of 3 sessions per week.
  Interventions: Other: Whole Body Vibration; Other: Aerobic Exercise

INTERVENTIONS:
Other: Whole Body Vibration — Each exercise session will be performed with a frequency of 30 Hz and an amplitude of 2 mm. Participants are in a 110° squat position on the platform (the degree will be adjusted using a goniometer). Participants will exercise for 16 minutes from week one to week three, 20 minutes from week four to week six and 24 minutes from week seven to week eight, respectively (8 iterations and 1 minute of vibration with 1 minute interval between each iteration)
  Arms: Whole Body Vibration
Other: Aerobic Exercise — From week one to week three, from week four to week six and from week seven to week eight, the participants will exercise for 30 minutes (5 minutes of running at 60-70% of heart rate and 5 minutes of active rest at 30-45% of maximum heart rate), 42 minutes (7 minutes of running at 60-70% of heart rate and 7 minutes of active rest at 30-45% of maximum heart rate) and 60 minutes (10 minutes of running at 60-70% of heart rate and 10 minutes of active rest at 30-45% of maximum heart rate). The exercise sessions consist of warm-up, main program and cool-down phases.

SUMMARY:
The aim of this interventional study is to investigate the effect of whole body vibration therapy on muscle oxygenation, vibration sensation, functional capacity and balance in individuals with Type 2 diabetes.

The main questions aimed to be answered are:

* Does whole body vibration therapy affect peripheral muscle oxygenation?
* Does whole body vibration therapy improve vibration sense, functional capacity and balance compared to aerobic exercise? Participants' muscle oxygenation, vibration sensation, functional capacity and balance parameters will be assessed. They will participate in a whole body vibration therapy or aerobic training program.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* Being diagnosed with type 2 diabetes
* 18 years of age or older
* HbA1c level to be 6.5-10%
* Having a clinical history of diabetes between 2-10 years
* Receiving oral hypoglycemic agent treatment
* At least three HbA1c measurements within 12 to 24 months
* Hemoglobin variability score (HVS) <50
* Being able to walk independently
* Mini mental test score ≥ 24
* Vastus lateralis muscle adipose tissue thickness <20mm
* BMI <30 kg/m2

Exclusion Criteria:

* Previous or concurrent psychiatric, neurological, orthopedic or systemic illness
* Use of insulin in treatment
* Diabetic neuropathy
* Foot ulcer
* Participation in any exercise program in the last 6 months
* History of major hypoglycemia in the last 12 months
* Working or have worked in a job with high exposure to mechanical whole body vibrations
* Conditions that may contraindicate whole body vibration (deep vein thrombosis, severe osteoporosis, active cancer, implanted medical devices, etc.)
* Hearing, vision and perception problems that may affect research results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Muscle Oxygenation | 8 weeks
  Vastus lateralis muscle oxygenation will be evaluated with Near-Infrared Spectroscopy at rest, during and after the 6-Minute Walk Test (6MWT)

SECONDARY OUTCOMES:
Vibration sense | 8 weeks
  The sense of vibration will be assessed with a 128 Hz diapason. The lower end of the device will be brought into contact with the plantar surface of the first metatarsal bone, the medial malleolus, and the medial tuberosity of the tuberositas tibia in both lower extremities of the individual. The moment the diapozone touches the tested areas will be considered as the zero-second (0th second, start), and the test will be terminated when the individual perceives that the vibration disappears completely and the time will be recorded in seconds. Three trials will be performed on the areas in both lower extremities, and the average will be reported.
The Timed Up & Go Test | 8 weeks
  It is a measurement that evaluates functional mobility, dynamic balance, fall risk and postural stability that can be applied for different purposes in different age and patient groups. The activities that make up the test evaluate the transition from sitting to standing position, walking, turning, and sitting again, which are necessary for functional mobility and dynamic balance. The TUG test measures the time it takes for an individual to get up from a standard chair with armrests and walk a distance of 3 meters, return from a designated or marked place, return to the chair, and sit back down.
The 6 minute walk test | 8 weeks
  The individual is asked to walk on a certain track for 6 minutes. The test is performed in a closed area, on a flat surface of 30 m in length and under the supervision of the evaluator. After six minutes, the total distance walked is recorded in meters.
The 30-second Chair Stand Test | 8 weeks
  In a chair with a sitting height of 43.2 cm and a back supported, the patient is asked to sit and stand as quickly as possible. The patient sits in the chair. They cross their hands on their chest. Before the test, 2 attempts are made. The number of sitting down times is noted by keeping a 30-second timer with a stopwatch. Less than 10 sit-ups in 30 seconds indicates lower extremity muscle weakness.
Balance | 8 weeks
  Balance assessment will be performed with the Biodex Balance System (Biodex Medical Systems Inc., Shirley, NY, USA). The static balance test (eyes open-closed) test, which measures the angular movement of the center of gravity, will be used in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Faculty of Health, Department of Physiotherapy and Rehabilitation, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No